CLINICAL TRIAL: NCT01788345
Title: Prospective Trial of the Bilevel Positive Airway Pressure (by Boussignac) in Emergency Department of Non-invasive Patients Presenting With Acute Hypercapnic Respiratory Failure
Acronym: Boussignac
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vygon GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 445-12
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Acute-on-chronic Respiratory Failure
Keywords: non-invasion ventilation; Boussignac
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- non-invasive ventilation (Experimental)
  Interventions: Other: non- invasive ventilation

INTERVENTIONS:
Other: non- invasive ventilation — non-invasive bi-level ventilation with IPAP and EPAP.
  Other Names: Boussignac

SUMMARY:
The purpose of this study is to determine whether the new Boussignac-system of non-invasive ventilation is as good as the conventional non-invasive System in patients presenting with acute hypercapnic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* 7,25 ≤ pH ≤ 7,35
* PaCO2 ≥ 45 mmHg

Exclusion Criteria:

* pH < 7,24
* incapable of collaboration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Sinking pCO2 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Budweiser, PD, Study Director
Locations (1):
- RoMed Klinikum Rosenheim, Rosenheim, Bavarian, Germany